CLINICAL TRIAL: NCT05311397
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of A166 in Patients With Unresectable, Locally Advanced or Metastatic HER2-expressing Solid Tumors (KL166-I-01-CTP)
Brief Title: A Study of A166 in Patients With Advanced Solid Malignant Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KL166-I-01-CTP
Record Dates: First submitted 2022-03-07; First posted 2022-04-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This 2-part, open-label, PhaseⅠstudy will administer A166 by IV infusion once every 3 weeks. Sequential dose-escalation cohorts are planned using a 3+3 design. An expansion study will be conducted based on the RS2D with comprehensive analysis of safety, tolerability, and pharmacokinetic data in the first phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first stage（Dose-escalation） (Experimental): According to the initial dose, the highest dose and the modified Fibonacci method, the dose escalation of A166 for injection is designed as: 0.1 mg/kg, 0.3 mg/kg, 0.6 mg/kg, 1.2 mg/kg, 2.4 mg/kg, 3.6 mg/kg, 4.8 mg/kg (the highest dose is tentatively set at 4.8 mg/kg).
  Interventions: Drug: A166
- The second stage（Dose-expansion） (Experimental): The administered dose of A166 for injection is RS2D obtained in the first stage .
  Interventions: Drug: A166

INTERVENTIONS:
Drug: A166 — A166 is an Antibody Drug Conjugate (ADC) targeting HER2 expressing cancer cells.

SUMMARY:
This is a single arm, open-label, dose-escalation and dose-expansion phase I study evaluating A166 in patients with HER2-expressing locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The first stage will determine the recommended stage 2 dose (RS2D) in patients with unresectable, locally advanced or metastatic HER2-expressing solid tumors based on safety, tolerability, pharmacokinetic characteristics and antitumor activity. The second stage will assess the safety, tolerability, pharmacokinetic characteristics and antitumor activity in dose-expansion cohorts (RS2D:3.6 mg/kg, 4.8 mg/kg and 6.0 mg/kg dose groups).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent form;
2. Age ≥ 18 years old, no gender limit;
3. Patients had a histologically confirmed incurable locally advanced or metastatic solid tumors;
4. Determined HER2-positive disease (detected by ISH or NGS) or HER2-expressing disease by evaluation or detection. Definition of HER2 expression in this study: Immunohistochemistry [IHC] ≥ 1＋;
5. Patients unable to benefit from the available standard treatment according to the judgment of the investigator;
6. White blood cell count (WBC) ≥ 4.0×109/L or ≥ lower limit of normal value; Neutrophil count (NEUT) ≥ 1.5×109/L; Platelet count (PLT) ≥ 100×109/L; Hemoglobin concentration ≥ 9.0 g/dL;
7. Total bilirubin (TBIL) ≤ 1.5×ULN. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN). For patients with liver metastases, ALT and AST ≤ 5 times ULN, and for patients with liver and/or bone metastases, alkaline phosphatase ≤ 5 times ULN;
8. Creatinine clearance rate ≥ 50 ml/min;
9. Patients had an Eastern Cooperative Oncology Group (ECOG)performance status of 0 or 1, the expected survival time is ≥ 3 months;
10. During the study period and within 7 months after the final administration of A166, patients with fertility (regardless of male and female) must receive effective medical contraceptive measures;
11. The patients must recover from all acute toxicities of the previous treatment (relieved to grade 1 or baseline), except for hair loss and vitiligo;

Exclusion Criteria:

1. Severe or uncontrollable heart disease requiring treatment, or grade 3 or 4 congestive heart failure according to the New York Society of Cardiology (NYHA), or unstable angina pectoris that cannot be controlled by drugs, or history of myocardial infarction within 6 months prior to enrollment, or severe arrhythmia requiring medical treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia);
2. History of ≥ Grade 3 allergic reaction to trastuzumab;
3. Permanent with drawal of trastuzumab due to any previous toxicity;
4. Patients with brain metastases who have symptoms or who have received the radiotherapy or surgery within 3 months before the first administration;
5. Patients requiring oxygen therapy in daily activities;
6. Grade 2 or higher peripheral neuropathy;
7. Any chemotherapy, hormone therapy (except dexamethasone), radiotherapy, immunotherapy or biological therapy received within 4 weeks before the first administration;
8. Prior-treatment with other clinical research drugs within 4 weeks before the first administration;
9. Patients who have undergone major surgery within 4 weeks before the first administration;
10. Active hepatitis B (hepatitis B surface antigen positive and HBV-DNA higher than the upper limit of reference value) or hepatitis C (positive hepatitis C virus antibody and HCV-RNA higher than the upper limit of reference value); current or past alcoholics ; Liver cirrhosis;
11. Known active human immunodeficiency virus (HIV);
12. Systemic diseases that cannot be controlled, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, glaucoma, etc according to investigator's judgment;
13. Current pregnancy or lactation;
14. QTc interval> 470 ms according to the baseline measurement:;
15. Left ventricular ejection fraction (LVEF) <45% according to the echocardiogram (ECHO) or multi-gate circuit controlled acquisition (MUGA) ;
16. Previous cumulative doxorubicin accumulation > 360 mg/m2 or its equivalent dose;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to RECIST v 1.1

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to 24 month
  From the date that response criteria are first met to the first occurrence of PD as determined by the investigators according to RECIST v1.1 or death from any cause, whichever occurs first
Progression-free survival(PFS) | up to 24 month
  PFS, defined as the active comparator arm frist dosing of A166 injection to the first occurrence of disease progression as determined by the investigators according to RECIST v1.1 or death from any cause, whichever occurs first
Overall Survival (OS) | up to 24 month
  OS, defined as the time from randomization to death or lose of follow, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No